CLINICAL TRIAL: NCT02561832
Title: A Phase I, Open-Label, 2 Part Multicentre Study to Assess the Safety, Tolerability and Efficacy of Olaparib in Combination With Carboplatin: Part A: Dose Escalation of Olaparib in Combination With Carboplatin in Patients With Advanced HER-2 Negative Breast Cancer; Followed by Part B: an Expansion Phase of Olaparib in Combination With Carboplatin in the Neoadjuvant Treatment of HER-2 Negative Breast Cancer Patients With Germline BRCA1/2 Mutations
Brief Title: A Phase I, Open-Label, 2 Part Multicentre Study to Assess the Safety and Efficacy of Olaparib in Combination With Carboplatin in Patients With Advanced HER-2 Negative Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This decision was based upon strategic considerations impacting the clinical development of olaparib in this indication.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D081EC00001
Record Dates: First submitted 2015-08-13; First posted 2015-09-28 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — olaparib; Carboplatin; Anthracyclines; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Part A: ascending doses of olaparib in combination with carboplatin will be administered to investigate safety and tolerability and to define the MTD and/or RD for part B. Patients will be treated with this combination up to cycle 4, after cycle 4 they can continue with combination or monotherapy (carboplatin or olaparib). Cohorts will be started sequentially, based on SRC recommendation. Part B will start after MTD/RD identification in part A. Patients will receive olaparib and carboplatin combination for first 4 cycles (21 days per cycle), at the dose, frequency and schedule recommended from Part A. This will be followed by another 4 cycles of standard cancer therapy consisting of anthracycline and cyclophosphamide regimen. Total of 8 treatment cycles will be given before final surgery
  Interventions: Drug: Olaparib; Drug: Carboplatin; Drug: Anthracycline; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Olaparib — tablets taken orally twice daily
Drug: Carboplatin — intravenous injections on day one of each cycle
Drug: Anthracycline — The choice of anthracycline and cyclophosphamide (AC) regimen in Part B will be up to local Investigator following international guidelines
Drug: Cyclophosphamide — The choice of anthracycline and cyclophosphamide (AC) regimen in Part B will be up to local Investigator following international guidelines

SUMMARY:
This is an open-label study to assess the safety, tolerability and efficacy of olaparib in combination with carboplatin. There are two parts in this study: Part A, a dose escalation in patients with advanced Human Epidermal Growth Factor 2 (HER-2) negative breast cancer and Part B, a dose expansion in the neoadjuvant treatment of HER-2 negative breast cancer patients with germline Breast Cancer Susceptibility Gene (BRCA)1/2 mutations.

DETAILED DESCRIPTION:
In Part A up to 36 evaluable patients with advanced breast cancer will be enrolled across 6 cohorts. The total number of patients will depend on the number of dose escalations necessary to enable a decision to be made on the recommended dose to take forward into Part B of the study.

The planned dose escalation will start with cohort 1, where patients will receive carboplatin (AUC5) on day 1 of cycle 1, and will start dosing with olaparib tablets at the dose of 50 mg twice daily (bd) on day 4 until day 19 of cycle 1 inclusive (a total of 16 days per cycle). Patients will receive carboplatin on day 1 of each 3 weeks cycle in combination with olaparib for a total of 4 cycles. Provided that there are no safety concerns after assessment of 6 evaluable patients in the first cohort, patients in subsequent cohorts may be dosed following Safety Review Committee (SRC) approval. Dose escalation scheme may be adjusted during the study on the basis of emerging safety, efficacy and pharmacokinetic data. Those patients in Part A who tolerate the combination up to and including cycle 4 may remain on treatment, either continuing with the combination, with carboplatin alone at the same AUC or with olaparib alone at the dose of 300 mg bd, if in the opinion of the treating Investigator, a patient is deemed to be deriving clinical benefit from treatment. In these cases, a patient may remain on treatment until progression, unacceptable toxicity or until other discontinuation criteria are met. Beyond cycle 4, patients will undergo assessments in line with the clinical protocol. Once the maximum tolerated dose (MTD) and/or recommended dose (RD) has been defined in Part A, a dose expansion phase, Part B will begin and this will include up to 21 patients with HER2 negative breast cancer, with a deleterious or suspected deleterious germlineBRCA1/2 (gBRCA1/2) mutation, who are deemed eligible for neoadjuvant therapy.

Part B will explore the safety, tolerability and efficacy of the combination of olaparib and carboplatin in terms of pathological complete response (pCR) rate. Neoadjuvant systemic therapy will consist of the following anti-cancer drugs for a total of 8 cycles of treatment:

* The first 4 cycles (cycle 1 to cycle 4: 12 weeks) will be based on combination of olaparib, at the defined RD and schedule from Part A, with carboplatin. It is expected that a cycle of treatment would be 3 weeks.
* Another 4 cycles (cycle 5 to cycle 8) will be based on a combination of an anthracycline and cyclophosphamide (AC). The choice of the AC regimen will be up to local Investigator following international guidelines (National Comprehensive Cancer Network (NCCN), European Society for Medical Oncology (ESMO), and St Gallen).

The tumour response will be assessed through careful clinical examination and also with radiological examinations between cycle 4 and 5 and at the end of neoadjuvant part, before surgery. Additionally, tumour biopsy will be performed within 7 days before cycle 5 day 1, after completion of carboplatin and olaparib combination therapy and early pathological response assessed by local pathologist. Curative-intent surgery should be performed following completion of neoadjuvant treatment in all patients, 3 to 5 weeks after day 1 of the last cycle of neoadjuvant treatment.

A decision has been made to stop recruitment after Part A cohort 2, and to not start Part B of the study. The protocol has been amended to define that the collection of clinical data will stop once the final patient from cohort 2 of Part A has completed 4 cycles or all patients from cohort 2 of Part A discontinue prior to end of cycle 4 to enable data analysis and reporting. The database would close at this time point, however AstraZeneca commits to providing study treatment to ongoing patients that continue to receive clinical benefit, in Investigator's judgment. Patients who remain on study treatment after this time point will be monitored according to routine clinical practice as defined by the Investigator and no clinical data will be collected, other than SAEs and drug dispensing/accountability.

ELIGIBILITY:
Inclusion criteria

* Male or female aged ≥18 years
* Normal organ and bone marrow function, measured within 28 days prior to administration of study treatment
* Eastern Cooperative Oncology Group performance status of 0-1
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential.

Additional for patients participating in Part A only

* Advanced or metastatic breast cancer that is HER-2 negative (HR positive or HR negative)
* Between 0 and 2 lines of prior cytotoxic chemotherapy. Additional for patients participating in Part B only
* Patients with operable breast adenocarcinoma and no evidence of metastatic disease are allowed.
* Patient must meet at least one of the following criteria: Clinical primary tumour size defined as T2 or above, clinical or patho-histological evidence of regional lymph nodes involvement (N+), grade 2-3 disease
* Availability of formalin fixed, paraffin embedded tumour sample from diagnostic biopsies (Not Applicable for patients at sites in Israel)
* Histological confirmation of HER-2 negative breast cancer
* Documented germline mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious
* Eligible for neo-adjuvant chemotherapy, but have not yet received neoadjuvant chemotherapy for breast cancer (chemo-naive) Exclusion criteria
* Exposure to an investigational product within 30 days or 5 half-lives (whichever is the longer) prior to enrolment
* Prior use of Poly ADP Ribose Polymerase (PARP) inhibitors
* Patients with a known hypersensitivity to olaparib or carboplatin
* Concurrent treatment with an ovarian hormonal replacement therapy or with hormonal agents such as raloxifene, tamoxifen or other selective estrogen receptor modulator. Patient must have discontinued use of such agents 3 weeks prior to beginning study treatment. Luteinising hormone-Releasing hormone (LHRH) analogues are allowed for all patients in Part A.
* Concomitant use of known potent Cytochrome P450 3A4 (CYP3A4) inhibitors and inducers
* Persistent toxicities (Common Terminology Criteria for Adverse Event (CTCAE) grade ≥2 and neuropathy CTCAE > grade 1) caused by previous cancer therapy, excluding alopecia - Patient with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML
* Patient must have recovered from any effects of any major surgery
* Patient considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled seizures or active uncontrolled infection
* Patient with known active Hepatitis B or C, or Human immunodeficiency virus (HIV)
* Other malignancy within the last 5 years (few exceptions apply). Additional for patients participating in Part A only
* Prior chemotherapy within 3 weeks of study entry
* Other anti-cancer therapy (eg, targeted biotherapy of hormonal agents) within 3 weeks of study entry
* Radiation therapy within 4 weeks or radionuclide treatment within 6 weeks of treatment start
* Prior use of platinum compound in the advanced or metastatic setting. Previous exposure to platinum compounds is allowed only if they were used in early adjuvant or neoadjuvant setting with relapse occurring >6 months after the last platinum administration and if there is no residual toxicity
* Patient with a history of treated Central Nervous System (CNS) metastases are eligible, provided they meet certain protocol-specified criteria.

Additional for patients participating in Part B only

* Prior treatment (local or systemic) of their breast tumour. Sentinel lymph node biopsy is considered as diagnostic procedure and therefore is authorized before neoadjuvant treatment in part B
* Patients with inflammatory breast cancer or patients with inoperable locally advanced breast cancer (including T4 lesions) at the time of enrolment.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Balmana, Principal Investigator — Hospital Vall d'Hebron, Barcelona, Spain; Tiffany Traina, Principal Investigator — Memorial Sloan Kettering Cancer Center, New York, USA
Locations (6):
- United States (2):
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Valencia
  - Research Site, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened between 06 November 2015 and 02 June 2016 at 7 medical centers in 2 countries
Pre-assignment Details: At screening, consenting patients were assessed to ensure that they met eligibility criteria. Once eligibility criteria were confirmed, patients underwent assessments applicable for the visit. Procedures that were part of standard of care may have occurred before informed consent was obtained.
Groups:
- Cohort 1: Olaparib 50mg, bid days 4 to 19 Carboplatin AUC5 on day 1 every 3 week
- Cohort 2: Olaparib 50mg, bid days 4 to 11 Carboplatin AUC5 on day 1 every 3 weeks
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 8 | 7
INFORMED CONSENT OBTAINED | 8 | 7
Completed (Subjects were still receiving study treatment when the study was terminated early by the Sponsor.) | 1 | 3
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Disease progression | 3 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)/Intention to treat (ITT): the primary statistical analysis of the efficacy of olaparib/carboplatin included all patients who signed the consent form, regardless of whether the treatment was actually received or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (14.57) | 47.7 (16.18) | 51.1 (15.15)
Age, Customized [Number; unit: Participants]
  >=18 to <33 | 0 | 1 | 1
  >=33 to <50 | 4 | 3 | 7
  >=50 to <65 | 1 | 2 | 3
  >=65 | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Subjects Reporting Adverse Events (AEs)
Description: Treatment-emergent AEs (TEAEs) defined as events occurring on or after cycle 1, day 1 up to and including 30 days after last dose (approximately 114 days).
Time Frame: From day 1 cycle 1, up to and including 30 days after last dose
Population: Safety analysis set consisting of all subjects who received at least one dose of study treatment
Measure: Number; unit: Participants
Groups:
- Cohort 1: Olaparib 50mg, bid days 4 to 19 Carboplatin AUC5 on day 1 every 3 weeks
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 7
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: AEs, including SAEs, were collected from time of signature of informed consent throughout the Treatment period (four 3-week cycles) up to and including the 30-day Follow-up period (approximately 142 days).
Description: All ongoing and any new AEs/SAEs identified during the 30-calendar day Follow-up period, after the last dose of study medication were required to be followed to resolution.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/7
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=7)
Anaemia (Blood and lymphatic system disorders) | 8 (10) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (10) | 3 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (10) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (10)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2)
Asthenia (General disorders) | 3 (3) | 2 (2)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (6) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (3)
Platelet count decreased (Investigations) | 3 (5) | 3 (5)
Weight decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to a small number of subjects analyzed (N=15).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No